CLINICAL TRIAL: NCT05437237
Title: Algorithm Development Through Artificial Intelligence for the Triage of Stroke Patients in the Ambulance With Electroencephalography
Brief Title: Algorithm Development Through AI for the Triage of Stroke Patients in the Ambulance With EEG
Acronym: AI-STROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jonathan Coutinho, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL75429.018.20
Record Dates: First submitted 2022-06-07; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry electrode cap EEG (Experimental): All patients that are included in the study will undergo a dry electrode electroencephalography (EEG).
  Interventions: Diagnostic Test: Dry electrode EEG

INTERVENTIONS:
Diagnostic Test: Dry electrode EEG — A single dry electrode electroencephalography (EEG) will be performed in each patient that is included in this study. For this purpose the Waveguard touch dry electrode EEG cap and compatible eego mini amplifier (ANT Neuro B.V., Hengelo, Netherlands) are used to record and amplify the EEG signal, respectively. Both products are CE marked as medical devices in the European Union and will be used within the intended use as described in the user manuals.

SUMMARY:
Endovascular thrombectomy (EVT) enormously improves the prognosis of patients with large vessel occlusion (LVO) stroke, but its effect is highly time-dependent. Direct presentation of patients with an LVO stroke to an EVT-capable hospital reduces onset-to-treatment time by 40-115 minutes and thereby improves clinical outcome. Electroencephalography (EEG) may be a suitable prehospital stroke triage instrument for identifying LVO stroke, as differences have been found between EEG recordings of patients with an LVO stroke and those of suspected acute ischemic stroke patients with a smaller or no vessel occlusion. The investigators expect EEG can be performed in less than five minutes in the prehospital setting using a dry electrode EEG cap. An automatic LVO-detection algorithm will be the key to reliable, simple and fast interpretation of EEG recordings by ambulance paramedics. The primary objective of this study is to develop one or more novel AI-based algorithms (the AI-STROKE algorithms) with optimal diagnostic accuracy for identification of LVO stroke in patients with a suspected acute ischemic stroke in the prehospital setting, based on ambulant EEG data.

DETAILED DESCRIPTION:
RATIONALE

Large vessel occlusion (LVO) stroke causes around 30% of acute ischemic strokes (AIS) and is associated with severe deficits and poor neurological outcomes. Endovascular thrombectomy (EVT) enormously improves the prognosis of patients with LVO stroke, but its effect is highly time-dependent. Because of its complexity and required resources, EVT can be performed in selected hospitals only. In the Netherlands, approximately half of the EVT-eligible patients are initially admitted to a hospital incapable of performing EVT, and - once it has been ascertained that the patient requires EVT - the patient needs to be transported a second time by ambulance to an EVT-capable hospital. Interhospital transfer leads to a treatment delay of 40-115 minutes, which decreases the absolute chance of a good outcome of the patient by 5-15%. To solve this issue, a prehospital stroke triage instrument is needed, which reliably identifies LVO stroke in the ambulance, so that these patients can be brought directly to an EVT-capable hospital. Electroencephalography (EEG) may be suitable for this purpose, since it shows almost instantaneous changes in response to cerebral blood flow reduction. Moreover, significant differences between EEGs of patients with an LVO stroke and those of suspected AIS patients with a smaller or no vessel occlusion have been found. A dry electrode EEG cap enables ambulance paramedics to perform an EEG in the prehospital setting, with significant reduced preparation time compared to conventional wet electrode EEG. An automatic LVO-detection algorithm will be the key to reliable, simple and fast interpretation of the EEG by paramedics, enabling direct admission of suspected AIS patients to the right hospital.

HYPOTHESIS

An EEG-based algorithm, developed with artificial intelligence (AI), will have sufficiently high diagnostic accuracy to be used by ambulance paramedics for prehospital LVO detection.

OBJECTIVE

The primary objective of this study is to develop one or more novel AI-based algorithms (the AI-STROKE algorithms) with optimal diagnostic accuracy for identification of LVO stroke in patients with a suspected AIS in the prehospital setting, based on ambulant EEG data.

STUDY DESIGN

AI-STROKE is an investigator-initiated, multicenter, diagnostic test accuracy study.

STUDY POPULATION

Part A: Adult patients with a (suspected) AIS, in the prehospital setting. Part B: Adult patients with a (suspected) AIS, in the in-hospital setting.

INTERVENTION

A single EEG measurement with a dry electrode cap (approximately 2 minutes recording duration) will be performed in each patient. In addition, clinical and radiological data will be collected. EEG data will be acquired with a CE approved portable dry electrode EEG device.

MAIN END POINTS

Primary end point: Based on the EEG data, and using the final diagnosis based on CT angiography data established by an adjudication committee as the gold standard, one or more novel AI-based EEG algorithms (the AI-STROKE algorithms) will be developed with maximal diagnostic accuracy (i.e. area under the receiver operating characteristic curve; AUC) to identify patients with an LVO stroke of the anterior circulation in a population of patients with suspected AIS.

Secondary end points:

* AUC, sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the AI-STROKE algorithms based on ambulant EEG for diagnosis of LVO of the anterior circulation in suspected AIS patients in the prehospital setting;
* AUC, sensitivity, specificity, PPV and NPV of existing EEG algorithms based on ambulant EEG for diagnosis of LVO stroke of the anterior circulation in suspected AIS patients in the prehospital setting;
* AUC, sensitivity, specificity, PPV and NPV of existing and newly developed EEG algorithms based on ambulant EEG for detection of LVO stroke of the posterior circulation, intracerebral hemorrhage, transient ischemic attack, and stroke mimics;
* Technical and logistical feasibility (e.g. in terms of EEG channel reliability) of paramedics performing ambulant EEG in patients with a suspected AIS in the prehospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Suspected AIS, as assessed by the attending ambulance paramedic, or a known LVO stroke;
* Onset of symptoms or last seen well < 24 hours before EEG acquisition;
* Age of 18 years or older;
* Written informed consent by patient or legal representative (deferred).

Exclusion Criteria:

* Skin defect or active infection of the scalp in the area of the electrode cap placement;
* (Suspected) COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1192 (Estimated)
Dates: Start 2022-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
One or more novel AI-based EEG algorithms based on dry electrode EEG-data with optimal diagnostic accuracy for LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  One or more novel artificial intelligence (AI) based electroencephalography (EEG) algorithms (the AI-STROKE algorithms) with maximal diagnostic accuracy to identify patients with an large vessel occlusion of the anterior circulation (LVO-a) in a population of patients with suspected acute ischemic stroke. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.

SECONDARY OUTCOMES:
AUC of the AI-STROKE algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Area under the receiver operating characteristic curve (AUC) of the AI-STROKE algorithms based on ambulant electroencephalography (EEG) for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
Sensitivity of the AI-STROKE algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Sensitivity of the AI-STROKE algorithms based on ambulant electroencephalography (EEG) for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
Specificity of the AI-STROKE algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Specificity of the AI-STROKE algorithms based on ambulant electroencephalography (EEG) for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
PPV of the AI-STROKE algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Positive predictive value (PPV) of the AI-STROKE algorithms based on ambulant electroencephalography (EEG) for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
NPV of the AI-STROKE algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Negative predictive value (NPV) of the AI-STROKE algorithms based on ambulant electroencephalography (EEG) for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
AUC of existing EEG algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Area under the receiver operating characteristic curve (AUC) of existing electroencephalography (EEG) algorithms based on ambulant EEG for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
Sensitivity of existing EEG algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Sensitivity of existing electroencephalography (EEG) algorithms based on ambulant EEG for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
Specificity of existing EEG algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Specificity of existing electroencephalography (EEG) algorithms based on ambulant EEG for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
PPV of existing EEG algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Positive predictive value (PPV) of existing electroencephalography (EEG) algorithms based on ambulant EEG for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
NPV of existing EEG algorithms for diagnosis of LVO-a | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Negative predictive value (NPV) of existing electroencephalography (EEG) algorithms based on ambulant EEG for diagnosis of large vessel occlusion of the anterior circulation (LVO-a) in suspected acute ischemic stroke patients in the prehospital setting. For each patient a single dry electrode electroencephalography (EEG) will be performed and the presence or absence of an LVO-a will be assessed based on CT angiography data acquired at the emergency department.
AUC of existing and newly developed EEG algorithms for detection of LVO-p, intracerebral hemorrhage, transient ischemic attack, and stroke mimics | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Area under the receiver operating characteristic curve (AUC) of existing and newly developed electroencephalography (EEG) algorithms based on ambulant EEG for detection of an large vessel occlusion of the posterior circulation (LVO-p), intracerebral hemorrhage, transient ischemic attack, and stroke mimics.
Sensitivity of existing and newly developed EEG algorithms for detection of LVO-p, intracerebral hemorrhage, transient ischemic attack, and stroke mimics | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Sensitivity of existing and newly developed electroencephalography (EEG) algorithms based on ambulant EEG for detection of an large vessel occlusion of the posterior circulation (LVO-p), intracerebral hemorrhage, transient ischemic attack, and stroke mimics.
Specificity of existing and newly developed EEG algorithms for detection of LVO-p, intracerebral hemorrhage, transient ischemic attack, and stroke mimics | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Specificity of existing and newly developed electroencephalography (EEG) algorithms based on ambulant EEG for detection of an large vessel occlusion of the posterior circulation (LVO-p), intracerebral hemorrhage, transient ischemic attack, and stroke mimics.
PPV of existing and newly developed EEG algorithms for detection of LVO-p, intracerebral hemorrhage, transient ischemic attack, and stroke mimics | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Positive predictive value (PPV) of existing and newly developed electroencephalography (EEG) algorithms based on ambulant EEG for detection of an large vessel occlusion of the posterior circulation (LVO-p), intracerebral hemorrhage, transient ischemic attack, and stroke mimics.
NPV of existing and newly developed EEG algorithms for detection of LVO-p, intracerebral hemorrhage, transient ischemic attack, and stroke mimics | EEG-data for development of the algorithm will be recorded within 24 hours after onset of symptoms or last seen well
  Negative predictive value (NPV) of existing and newly developed electroencephalography (EEG) algorithms based on ambulant EEG for detection of an large vessel occlusion of the posterior circulation (LVO-p), intracerebral hemorrhage, transient ischemic attack, and stroke mimics.
Technical feasibility of performing ambulant EEGs in the prehospital setting | Feedback on technical issues by the paramedic that performs the EEG and by the EEG-expert, will be collected directly at arrival in the emergency department (within 24 hours after the patient is included in the study)
  Assessing whether it is technically possible for paramedics to perform ambulant electroencephalography (EEG) in patients with a suspected AIS in the prehospital setting.
Logistical feasibility of performing ambulant EEGs in the prehospital setting | Feedback on logistical issues by the paramedic that performs the EEG, will be collected directly at arrival in the emergency department (within 24 hours after the patient is included in the study)
  Assessing whether it is logistically possible for paramedics to perform ambulant electroencephalography (EEG) in patients with a suspected AIS in the prehospital setting.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Coutinho, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam University Medical Centers, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT05437237/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT05437237/ICF_001.pdf